CLINICAL TRIAL: NCT00916799
Title: VISN 23 COPD Case Management Using Home Telehealth Equipment
Brief Title: VISN 23 Chronic Obstructive Pulmonary Disease (COPD) Case Management Using Home Telehealth Equipment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Naresh A. Dewan, M.D., VA Nebraska Western Iowa Heathcare System, Omaha
Organization: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 00576
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: COPD
Keywords: telehealth; oximetry; copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oximeter arm and non-oximetry arm (Experimental)
  Interventions: Device: Use of Telehealth equipment (Viterian V-100)

INTERVENTIONS:
Device: Use of Telehealth equipment (Viterian V-100) — Patient will daily enter answers to questions generated from a home telehealth monitor
  Other Names: Viterian V-100

SUMMARY:
Looking at the use of home telehealth equipment and it's place in self management and education in patients who suffer moderate to severe Chronic Obstructive Pulmonary Disease (COPD). The patients in this group would be those patients who traditionally suffer from emphysema, and/or chronic bronchitis.

DETAILED DESCRIPTION:
Patients who have been admitted to the hospital, or who have frequent urgent care visits, who also suffer from COPD exacerbations will be given a home monitoring system. Daily, the patient will respond to a series of questions. The results of the question answers will be remotely monitored by a nurse case manager.

The objective is to measure compliance, resource use, and the ability for early recognition of an exacerbation of their COPD, and early implementation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* One or more hospital admissions or emergency room visits in last 2 Years.
* Patient must meet the VA home telehealth guideline that the patient is determined to be at high risk for poor clinical outcomes or increased unplanned health care utilization based on disease specific criteria and/or determined by physician provider

Exclusion Criteria:

* Any unstable medical condition that the investigator thinks would preclude effective participation in the study, or which would be expected to reduce life expectancy to less than 1 year.
* Unwilling or unable to provide consent
* Uncooperative or combative
* Does not have a compatible phone line
* Inability to use home telemedicine equipment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-11 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Patient compliance with utilizing home telehealth monitoring equipment in the two patient groups | six months
The amount of Home telehealth case management time utilized to provide patient monitoring in the two patient groups | six months

SECONDARY OUTCOMES:
Patient satisfaction The role of finger oximetry in the identification of exacerbations Number of hospitalizations and urgent care visits and how they relate to the use of home telehealth equipment | six months
Evaluate patient ease of using the home telehealth equipment in the two patient groups. | six months
Patient satisfaction in managing their disease in the two patient groups | six months
The number of COPD exacerbations, urgent care visits, and hospitalizations related to COPD in the two patient groups | six months
Correlate the effect of oxygen saturation monitoring on the early identification of COPD exacerbations | six months

CONTACTS AND LOCATIONS:
Overall Officials: Naresh A Dewan, M.D., Principal Investigator — VA Nebraska Western Iowa Healthcare System, Omaha
Locations (2):
- United States (2):
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Nebraska Western Iowa Healthcare System, Omaha, Omaha, Nebraska

REFERENCES:
- [Result] Noel HC, Vogel DC, Erdos JJ, Cornwall D, Levin F. Home telehealth reduces healthcare costs. Telemed J E Health. 2004 Summer;10(2):170-83. doi: 10.1089/tmj.2004.10.170. PMID 15319047
- [Result] Vontetsianos T, Giovas P, Katsaras T, Rigopoulou A, Mpirmpa G, Giaboudakis P, Koyrelea S, Kontopyrgias G, Tsoulkas B. Telemedicine-assisted home support for patients with advanced chronic obstructive pulmonary disease: preliminary results after nine-month follow-up. J Telemed Telecare. 2005;11 Suppl 1:86-8. doi: 10.1258/1357633054461697. PMID 16036007
- [Result] Rahimpour M, Lovell NH, Celler BG, McCormick J. Patients' perceptions of a home telecare system. Int J Med Inform. 2008 Jul;77(7):486-98. doi: 10.1016/j.ijmedinf.2007.10.006. Epub 2007 Nov 26. PMID 18023610